CLINICAL TRIAL: NCT02538003
Title: A Randomized, Open-label, Single Dose, Crossover, Phase Ⅰ Trial to Evaluate the Effect of Food on the Pharmacokinetics of LCB01-0371 in Healthy Male Subjects
Brief Title: To Evaluate the Effect of Food on Pharmacokinetics(PK), Phase I Clinical Study of LCB01-0371
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-13-1-03
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — delpazolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1(RT):LCB01-0371 Tablet 800mg (Experimental): 1. Period:LCB01-0371 Tablet 800mg(Reference: Taken drug before meal)
  2. Period: LCB01-0371 Tablet 800 mg(Test: Taken drug after meal)
  Interventions: Drug: LCB01-0371 Tablet 800 mg(R); Drug: LCB01-0371 Tablet 800 mg(T)
- Group 2(TR):LCB01-0371 Tablet 800mg (Experimental): 1. Period:LCB01-0371 Tablet 800mg(Test:taken drug after meal)
  2. Period: LCB01-0371 Tablet 800 mg(Reference:taken drug before meal)
  Interventions: Drug: LCB01-0371 Tablet 800 mg(R); Drug: LCB01-0371 Tablet 800 mg(T)

INTERVENTIONS:
Drug: LCB01-0371 Tablet 800 mg(R) — Reference: taken drug before meal
  Other Names: LCB01-0371 Tablet 400 mg 2 Tablet
Drug: LCB01-0371 Tablet 800 mg(T) — Test: taken drug after meal
  Other Names: LCB01-0371 Tablet 400 mg 2 Tablet

SUMMARY:
The purpose of this study is to assess safety, tolerability of LCB01-0371 after fasting/non-fasting food taken in healthy male subjects.

DETAILED DESCRIPTION:
A Randomized, Open-label, Single dose, Crossover, Phase Ⅰ Trial to evaluate the effect of food on the pharmacokinetics of LCB01-0371 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male between 20 and 40 years of age at the time of screening with body mass index (BMI) between 19 kg/m2 and 28 kg/m2 at the time of screening
2. Appropriated for a medical examination by interview,Vital sign,physical examination, local laboratory test result and 12-lead ECG
3. Capable of performing follow up visit, blood sampling
4. Agree to continue to use a medically reliable dual contraception and not to donate sperm in this protocol for the duration of the study and for 28 days after last dose of investigational product
5. Capable of giving written informed consent, willing to participate in this clinical trial, and willing to comply with all study requirements

Exclusion Criteria:

1. History of clinically significant disease such as digestive system, respiratory, musculoskeletal, cardiovascular, endocrine, neuropsychiatry, hematology, cardiovascular system
2. History of gastrointestinal problem (e.g. Crohn's disease, gastro-intestinal ulcer) within 180 days possibly affecting absorption of clinical trial drugs, or history of surgery (except simple appendectomy and herniotomy)
3. History of hypersensitivity reaction or history of clinically significant hypersensitivity reaction to LCB01-0371 or same class of the study drugs (linezolid) or other drugs including aspirin and antibiotics(except non active allergic rhinitis)
4. History of drug abuse or positive result at urine drug screening test at screening visit
5. Intake drug which expected to chronic influence of drug absorption or elimination within 30 days prior to screening visit
6. Other: Patients considered unable perform for the study by the investigator concerning

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | From date of randomization until follow up after 7 days from last hospital discharge

SECONDARY OUTCOMES:
Pharmacokinetics: AUClast(Area under the plasma concentration) | 0(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24hours
Pharmacokinetics: Cmax(Peak plasma concentration) | 0(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyong Chung, M.D., Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Bundang, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No